CLINICAL TRIAL: NCT05366205
Title: Prospective, Randomized Controlled Study on Immune Function Regulation by Strengthening Early Oral Nutritional Supplementation in Elderly Patients With Mild to Moderate COVID-19 on Hemodialysis
Brief Title: Immune Function in Elderly Patients With Mild to Moderate COVID-19 on Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, SHI YONGMEI, associate chief physician, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJYY01
Record Dates: First submitted 2022-04-30; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Hemodiafiltration
Keywords: COVID-19; Hemodiafiltration; immune function; Oral nutritional supplement
MeSH Terms: conditions — COVID-19 | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral nutritional supplements (Experimental): Patients in this arm will receive oral nutritional supplements 24-48 hours after admission，which is enteral nutrition emulsion(TPF-T).
  Interventions: Dietary Supplement: Oral nutritional supplement
- nutrition consultation (Sham Comparator): Patients in this arm will receive nutrition consultation was given in addition to basic treatment.
  Interventions: Behavioral: Nutrition consultation

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement — Enteral nutritional emulsion(TPF-T) will be given by oral intake,400ml per day, lasting for 7-10 days.
  Arms: Oral nutritional supplements
Behavioral: Nutrition consultation — Nutritional treatment advice will be given
  Arms: nutrition consultation

SUMMARY:
This randomized controlled trial will focus on the effects of early oral nutritional supplementation on immune function in elderly patients with mild to moderate COVID-19 on maintenance hemodialysis. The purpose of this study is to determine whether early oral nutritional supplementation can improve immune function and clinical outcomes.

DETAILED DESCRIPTION:
COVID-19 is in the midst of a global pandemic. Elderly patients are often susceptible and at high risk. Elderly patients on maintenance hemodialysis are often accompanied by a variety of complications, malnutrition is a common complication with an incidence of 23-73%. Due to a variety of risk factors, COVID-19 infection tends to develop into severe disease, and it takes longer for nucleic acid to turn negative.

This randomized controlled trial will focus on the effects of early oral nutritional supplementation on immune function in elderly patients with mild to moderate COVID-19 on maintenance hemodialysis. The purpose of this study is to determine whether early oral nutritional supplementation can improve immune function and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 and above;
2. Patients receiving hemodialysis with clinically confirmed end-stage renal disease
3. Positive diagnosis of COVID-19 by RT-PCR nasopharyngeal swab was classified as mild or moderate type
4. Patients who can eat on their own;
5. Patients had good compliance, fully understood the study content and signed informed consent.

Exclusion Criteria:

1. Contraindications of oral nutritional supplementation, such as intestinal obstruction and intestinal ischemia.
2. In an unstable state of vital signs such as shock.
3. In acute pancreatitis, cholecystitis acute attack period and 3 months after the last attack
4. Patients with moderate to severe cognitive impairment or mental diseases;
5. People who are allergic to intestinal nutrients
6. Refuse oral nutritional supplements

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
CD4 lymphocyte counts | Baseline to discharge date, an average of 3 weeks
lymphocyte count | Baseline to discharge date, an average of 3 weeks
T-lymphocyte subsets | Baseline to discharge date, an average of 3 weeks
  CD3+, CD4+, CD8+

SECONDARY OUTCOMES:
Change in body weight | Baseline to discharge date, an average of 3 weeks
change in white blood cell count | Baseline to discharge date, an average of 3 weeks
change in hemoglobin | Baseline to discharge date, an average of 3 weeks
change in albumin | Baseline to discharge date, an average of 3 weeks
change in C-Reactive Protein | Baseline to discharge date, an average of 3 weeks
change in procalcitonin | Baseline to discharge date, an average of 3 weeks
change in nutritional risk screening 2002(NRS 2002) score | Baseline to discharge date, an average of 3 weeks
  Scores range from 0 to 7，a score greater than or equal to 3 indicates nutritional risk
change in mini nutritional assessment short-form（MNA- SF） score | Baseline to discharge date, an average of 3 weeks
  Scores range from 0 to 14，a score of 0 to 7 indicates malnutrition，8-11 indicates risk of malnutrition, 12-14 indicates normal nutrition
change in Geriatric nutritional risk index(GNRI) score | Baseline to discharge date, an average of 3 weeks
  Higher scores mean a worse outcome
Length of hospital stay | Baseline to discharge date, an average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Shi, MD, Study Chair — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No